CLINICAL TRIAL: NCT04890340
Title: An International Multicenter Blind Comparative Controlled in Vitro Study of the Liquid Biopsy Test System of the Diagnostic Value, in Women With Various Forms of Breast Cancer in Comparison With Other Early Diagnostic Methods (Mammography/Ultrasound/MRI).
Brief Title: In Vitro Study of the Liquid Biopsy Test System of the Diagnostic Value, in Women With Various Forms of Breast Cancer
Acronym: ARNABreast
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ARNA Genomics US Inc. (Industry)
Collaborators: BIOMARKER-RU (Unknown)
Responsible Party: Sponsor
Other Study IDs: ARNA Breast 2021
Record Dates: First submitted 2021-04-19; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ARNA technology in general and the ARNA Breast test in particular are performed in a specialized laboratory. The courier service ships whole blood from the Clinic to the Laboratory. Thus, direct contact of the patient with the reagents does not occur, which increases the safety of the system. Plasma will be isolated from the sample in the Laboratory. Plasma is processed with a set of reagents, including inorganic and organic solutions and sets of specially synthesized biological components (oligonucleotides), for real-time polymerase chain reaction (RT-PCR) to determine the content of DNA fragments of selected oncological genes in a woman's blood plasma. The remaining plasma will be kept frozen for retests upon request. Samples will be not transferred to other countries.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women in age 35 to 65 with suspected breast cancer: Women in age 35 to 65 with suspected breast cancer, previously untreated. Additionally, eligible patients should have appropriate mammography results, either breast ultrasound or breast MRI.
  Interventions: Diagnostic Test: ARNA Breast
- Healthy Volunteers: Healthy woman in age 35 to 65.
  Interventions: Diagnostic Test: ARNA Breast

INTERVENTIONS:
Diagnostic Test: ARNA Breast — Women of the required age group, in case of suspicion of breast cancer, are sent to clarify the diagnosis for mammography or ultrasound of the mammary glands, or MRI. Based on the results of these studies, a biopsy is prescribed to make a final diagnosis. Before a biopsy to diagnose the presence / absence of breast cancer, patients do the blood sampling one time. The blood is processed in the Sponsor's laboratory. The test results are compared with the data obtained from the biopsy. The evaluation of the effectiveness of the method will be determined on the basis of the obtained data on the sensitivity and specificity of the test in relation to the reference method

SUMMARY:
The Study Objective is to evaluate the diagnostic efficacy of the liquid biopsy system versus the gold standard mammography (or MRI, or Ultrasound) diagnosis in patients with suspected breast cancer.

DETAILED DESCRIPTION:
Women of the required age group, in case of suspicion of breast cancer, are sent to clarify the diagnosis for mammography or ultrasound of the mammary glands, or MRI. Based on the results of these studies, a biopsy is prescribed to make a final diagnosis. Before a biopsy to diagnose the presence / absence of breast cancer, patients do the blood sampling one time. The blood is processed in the Sponsor's laboratory. The test results are compared with the data obtained from the biopsy. The evaluation of the effectiveness of the method will be determined on the basis of the obtained data on the sensitivity and specificity of the test in relation to the reference method.

ELIGIBILITY:
Inclusion Criteria:

* Availability of signed and dated informed consent.
* Women from 35 to 65 years old, who are generally healthy, with suspected breast cancer. Or without suspicion of (control group)
* Presence of a documented referral diagnosis of "breast cancer"
* Presence of a documented biopsy referral
* Presence of mammography, ultrasound or MRI of the mammary glands no later than three months.

Exclusion Criteria:

* Pregnancy.
* Any other cancers diagnosed now or previously, with the exception of breast cancer.
* Therapy with cytostatics during the last three months.
* Chemotherapy within the past three months.
* Therapy with hormonal drugs, including all forms of contraceptive drugs.
* Therapy with other prohibited groups of drugs.
* Systolic blood pressure > 180 mm Hg. and / or diastolic blood pressure > 120 mm Hg. with repeated measurements.
* Simultaneous participation in another clinical study.
* Relative affiliation to the clinic, for example, the patient is a close relative of the researcher or a dependent person (for example, a clinic employee or student or a sponsor employee).
* A clinically significant condition or laboratory result that, in the opinion of the investigator, threatens the safety of the test subject, may interfere with assessments, or prevent the completion of the study.
* Failure to cooperate to participate in planned procedures, including the following examples: lack of understanding of language, mental illness, inability to visit the clinic.
* Diseases or conditions that may affect the conduct of the study or the interpretation of the results.
* History of organ transplantation.
* Blood transfusions within the last 6 months.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women of the required age group, in case of suspicion of breast cancer, are sent to clarify the diagnosis for mammography or ultrasound of the mammary glands, or MRI but before biopsy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-21 (Estimated); Primary Completion 2021-11-29 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of woman with positive ARNA Breast test confirmed by biopsy (Sensitivity) | through study completion, an average of 1 year
  Primary Measured Values for Efficiency Assessment:
  1. the absolute total number of matches between the results of the test system and mammography based on histological confirmation of the diagnosis;
  2. the sensitivity of the test by groups, particularly: the ratio of the number of true-positive test results to the total number of patients in the group with the presence of a character;
  3. the specificity of the test by groups, particularly: the ratio of the number of true-negative test results to the total number of patients in the group with no character. A group of samples from patients with a confirmed diagnosis of breast cancer will be divided into 4 subgroups depending on the biological subtype of cancer identified on the basis of IHC analysis (luminal A, luminal B, HER2/neu, triple negative), also for the subgroups obtained the primary measured values will be calculated to identify these quantities based on the biological subtype of breast cancer.

SECONDARY OUTCOMES:
Efficiency Evaluation | through study completion, an average of 1 year
  Estimation of the area under ROC-curve (AUC)
Relationship between test results and the age | through study completion, an average of 1 year
  Determination of a statistically significant relationship between test results and the age of patients at the time of testing
Positive predictive value | through study completion, an average of 1 year
  The ratio of true-positive test results to the total number of positive test results h) the ratio of true negative test results to the total number of negative test results (negative predictive value) i) Positive and negative likelihood ratio
Negative predictive value | through study completion, an average of 1 year
  The ratio of true negative test results to the total number of negative test results

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Tarabarov, MD, Study Director — BIOMARKER-RU

IPD SHARING:
Plan to Share IPD: No